CLINICAL TRIAL: NCT00382148
Title: A Phase IIb, Open-Label Study of Xolair (Omalizumab) in Peanut-Allergic Subjects Randomized to Study Drug in Study Q2788g (TOPS)
Brief Title: A Study of Xolair in Peanut-Allergic Subjects Previously Enrolled in Study Q2788g
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Q3623g
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2009-12-15 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-11

CONDITIONS: Peanut Hypersensitivity
Keywords: TOPS; Peanut allergy; Peanut-induced allergy; Allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity | interventions — Omalizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: omalizumab

INTERVENTIONS:
Drug: omalizumab — SC repeating dose

SUMMARY:
This is a Phase IIb, multicenter, open-label study available to active (Xolair) and control (placebo) subjects who have completed their final visit (or early termination visit, if applicable) for Study Q2788g, who meet the eligibility criteria of this study, and who provide consent to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Completion of last visit (or early termination visit, if applicable) for Study Q2788g
* Signed Informed Consent Form
* Use of an effective method of contraception for females of childbearing potential
* Body weight ≥ 20 kg and ≤ 150 kg
* IgE level ≤ 1300 IU/mL (Note: Subjects with an IgE < 30 IU/mL will be dosed at the lowest level on the dosing table [30 IU/mL], thus enabling better understanding of the role of Xolair in peanut allergic subjects who have low total IgE levels.)

Exclusion Criteria:

* Withdrawal from Study Q2788g prior to study closure or the final study visit (Week 36)
* Current participation in another investigational study
* Pregnancy or lactation
* History of brittle asthma
* Aspirin-sensitive asthma
* Known hypersensitivity to any ingredients of Xolair, including its excipients (sucrose, histidine, polysorbate 20)
* Have a polymorrphonuclear count <1500/uL
* Use of anti-coagulants, such as warfarin (Coumadin(R)), thrombolytic enzymes, or ticlopidine
* Current diagnosis of cancer, current investigation for possible cancer, or history of cancer (not including non-melanoma skin cancer)
* Thrombocytopenia as evidenced by a platelet count < 100,000/uL
* Any systemic condition requiring regular administration of an immunoglobulin

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wong, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab (Placebo in Q2788g); Omalizumab (Omalizumab in Q2788g): Either a minimum of 0.016 mg/kg/IgE (IU/mL) every 4 weeks or 0.008 mg/kg/IgE (IU/mL) every 2 weeks (based on dosing table)
Period: Overall Study
Arm/Group | Omalizumab (Placebo in Q2788g) | Omalizumab (Omalizumab in Q2788g)
Started | 4 | 7
Completed | 3 | 7
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab (Placebo in Q2788g) | Omalizumab (Omalizumab in Q2788g) | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Customized [Number; unit: participants] — Safety-analysis population
  participants
    6 to < 12 | 0 | 2 | 2
    >= 12 | 4 | 5 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 32.0 (23.5) | 17.3 (8.9) | 22.6 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: All grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0. An SAE is defined as an adverse event that results in death, is life threatening, requires hospitalization, results in significant disability, results in birth defect, or is considered a significant medical event by the investigator
Time Frame: Through Week 52
Population: Safety-analysis population
Measure: Number; unit: participants
Arm/Group | Omalizumab (Placebo in Q2788g) | Omalizumab (Omalizumab in Q2788g)
Number analyzed (Participants) | 4 | 7
participants
  Overdose | 0 | 1
  Depression | 0 | 1

2. Secondary Outcome: Food Allergen Exposure, Assessed on Patient-reported Questionnaire
Description: Participants were asked to record every 4 weeks in the food-related allergic event questionnaire: "Whether you were exposed to peanut, tree nut (cashew, almond, etc.), shellfish (shrimp, crab, etc.), eggs, milk, or other (please specify)" and "Did you have a reaction? (Yes/No)."
Time Frame: Every 4 weeks through Week 52
Measure: Number; unit: participants
Arm/Group | Omalizumab (Placebo in Q2788g) | Omalizumab (Omalizumab in Q2788g)
Number analyzed (Participants) | 4 | 7
participants
  Peanut | 1 | 3

3. Secondary Outcome: Food-allergic Reactions As Assessed by the Ewan Scale
Description: The Ewan scale has five ascending grades of severity from "Grade 1" to "Grade 5" (as well, there is a possible value of "Not Applicable"). Following a report of an allergic reaction to food on a patient-reported questionnaire, the reaction is graded by the study coordinator or Principle Investigator
Time Frame: Through Week 52
Population: safety-evaluable population
Measure: Number; unit: participants
Arm/Group | Omalizumab (Placebo in Q2788g) | Omalizumab (Omalizumab in Q2788g)
Number analyzed (Participants) | 4 | 7
participants
  Grade 1 | 0 | 1
  Grade 2 | 0 | 0
  Grade 3 | 1 | 2
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

4. Secondary Outcome: Nonserious Food-related Adverse Events (AEs) and Other Nonserious AEs
Description: All grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0. All AEs that do not meet any of the criteria for serious should be regarded as nonserious AEs.
Time Frame: Through Week 52
Population: safety-evaluable population
Measure: Number; unit: participants
Arm/Group | Omalizumab (Placebo in Q2788g) | Omalizumab (Omalizumab in Q2788g)
Number analyzed (Participants) | 4 | 7
participants
  Lymphadenopathy | 0 | 1
  Motion Sickness | 0 | 1
  Tinnitus | 0 | 1
  Diarrhoea | 0 | 2
  Abdominal Pain | 0 | 2
  Nausea | 0 | 2
  Vomiting | 0 | 1
  Lip Swelling | 0 | 1
  Oral Pruritis | 0 | 1
  Pyrexia | 0 | 2
  Injection Site Bruising | 1 | 1
  Fatigue | 0 | 1
  Nasopharyngitis | 0 | 2
  Laryngitis | 0 | 1
  Sinusitis | 0 | 1
  Upper Respiratory Tract Infection | 1 | 0
  Pharyngitis Streptococcal | 1 | 1
  Gastroenteritis | 0 | 1
  Otitis Media | 0 | 1
  Localised Infection | 0 | 1
  Anorexia | 0 | 1
  Arthralgia | 1 | 0
  Loss of Consciousness | 0 | 1
  Headache | 0 | 1
  Migraine | 0 | 1
  Dizziness | 0 | 1
  Hypoaesthesia | 0 | 1
  Menstruation Irregular | 1 | 0
  Cough | 0 | 3
  Nasal Congestion | 0 | 2
  Rhinitis Allergic | 1 | 0
  Asthma | 0 | 2
  Pharyngolaryngeal Pain | 0 | 2
  Rhinorrhoea | 0 | 1
  Throat Irritation | 0 | 1
  Eczema | 1 | 1
  Rash | 0 | 1

ADVERSE EVENTS:
Arm/Group | Omalizumab (Placebo in Q2788g) | Omalizumab (Omalizumab in Q2788g)
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/7
Other Adverse Events (participants affected / at risk) | 3/4 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (Placebo in Q2788g) (N=4) | Omalizumab (Omalizumab in Q2788g) (N=7)
Depression (Psychiatric disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (Placebo in Q2788g) (N=4) | Omalizumab (Omalizumab in Q2788g) (N=7)
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Injection Site Bruising (General disorders) | 1 | 1
Laryngitis (General disorders) | 0 | 1
Lip Swelling (Gastrointestinal disorders) | 0 | 1
Localised Infection (Infections and infestations) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Menstruation Irregular (Reproductive system and breast disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Motion Sickness (Ear and labyrinth disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Oral Pruritis (Gastrointestinal disorders) | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1
Pharyngitis Streptococcal (Infections and infestations) | 1 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study.